CLINICAL TRIAL: NCT05167201
Title: Does Domiciliary Nasal High Flow (NHF) Therapy Improve Patient Outcomes in Chronic Hypercapnic Respiratory Failure (CHRF) in the United Kingdom (UK): A Pre and Post Interventional Study
Brief Title: Domiciliary Nasal High Flow and Patient Outcomes in Chronic Hypercapnic Respiratory Failure in the United Kingdom
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Fisher and Paykel Healthcare (Industry); Royal Free Charity (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307348
Record Dates: First submitted 2021-11-01; First posted 2021-12-22 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Chronic Hypercapnic Respiratory Failure; Chronic Obstructive Pulmonary Disease; Obesity Hypoventilation Syndrome (OHS); Nasal High Flow; Health-related Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Intervention Model Description: Single arm pre and post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal High Flow (Experimental): The Nasal High Flow device is an integrated flow generator that delivers warmed and humidified air to spontaneously breathing patients through a variety of patient interfaces.
  Flow rates up to 60 litres/minute are available to the user, depending on the patient interface and mode of operation.
  Interventions: Device: Nasal High Flow

INTERVENTIONS:
Device: Nasal High Flow — High flow nasal cannula (NHF) is a device that delivers warmed and humid air through a high air flow rate, through the nose. It is used as a non-invasive ventilatory approach, which is relatively comfortable, in the management of respiratory failure and has been investigated in several studies evaluating the outcomes as domiciliary treatment in patients with COPD.

SUMMARY:
Chronic hypercapnic respiratory failure (CHRF) in the context of Chronic Obstructive Pulmonary Disease (COPD) and Obesity Hypoventilation Syndrome (OHS) is associated with increased mortality. The availability and effectiveness of domiciliary Non-invasive ventilation (NIV) treatment (when indicated) is key as this treatment can improve quality of life and reduce health-care costs from associated burden of disease. The emerging obesity epidemic means that there is now increased home mechanical ventilation set-ups in patients with obesity related respiratory failure (ORRF), yet there are no alternative treatments for patients struggling with domiciliary NIV.

Domiciliary NHF has been shown to improve health related quality of life in stable CHRF in patients with COPD and improve cost effectiveness yet there are no current studies looking at the use of domiciliary NHF and its outcomes in ORRF.

The study aims to deliver a pre and post intervention study evaluating patient reported and clinical outcomes in patients using NHF over twelve weeks, who have either COPD or OHS and have been unable to use domiciliary NIV. The study wishes to address key outcomes such as quality of life, clinical effectiveness, compliance and acceptability with the use of domiciliary NHF in both of these patient populations.

DETAILED DESCRIPTION:
This study is an investigator-initiated, unblinded, multi-centre, one arm pre and post interventional study evaluating the use of nasal high flow over twelve weeks, upon self-reported quality of life in adults aged 18 and above, with COPD or OHS and CHRF. This is not a comparator trial and will provide preliminary information on the intervention in a group of individuals who cannot comply with current guideline recommended therapy (with all strategies used to address any barriers to current treatment usage).

This study will therefore aim to evaluate if this treatment offers effective outcomes in this difficult to treat population thus reflecting the variations in practice and choices that occur for this group of individuals in real practice.

Ethical approval will be obtained from the research ethical committee of Brighton and Sussex. Informed consent will be obtained from all willing participants.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with chronic obstructive pulmonary disease (COPD) who meet these criteria for domiciliary NIV:

   - Diagnosis of COPD based on spirometry; The ration of the forced expiratory volume in the first one second (FEV1) to the forced vital capacity (FVC) of the lungs (FEV1/FVC ratio), of ⩽ 0.70

   And either of:
   * i) Recent inpatient admission with acute hypercapnic respiratory failure with persistent hypercapnia (pH ≥ 7.35 and PaCO2 ≥ 6 kilopascal (kPa)) 2-4 weeks after the acute episode or
   * ii) COPD with evidence nocturnal hypoventilation (sleep study demonstrating time under 90% saturations for 30% of the sleep time) or
   * iii) Stable CHRF (paO2 ⩽ 8 kPa and paCO2 ≥ 6 kPa)

   OR
2. All patients with OHS who meet these criteria for domiciliary NIV i) Diagnosis of OHS based on Body Mass Index > 30 kg/m2, daytime hypercapnia (PaCO2 ≥ 6kPa) and significant nocturnal hypoventilation (saturations ⩽ 90% for 30% of the total sleep time) or ii) Inpatient admission with acute hypercapnic respiratory failure requiring NIV referred for consideration of domiciliary treatment

who have been offered treatment with NIV and have:

3)

* discontinued or demonstrated poor compliance with domiciliary NIV (defined as ⩽ 4 hours usage for 70% of the nights at 4 months with all reasonable measures taken to address barriers to treatment use)
* evidence of sleep disordered breathing on a sleep study
* over or equal to 18 years of age
* able to provide informed consent
* able to participate for the duration of the study
* have an expected survival for greater than three months

All patients must meet inclusion criteria for 1 or 2 and all of 3

Exclusion Criteria:

* Unstable psychiatric disease
* Unable to return for review appointments e.g due to move home or lives a long distance from the study site
* Pregnancy
* Receiving home NIV treatment at time of inclusion to study
* Receiving home NIV treatment for other medical illnesses, for example neuromuscular disease
* Unable to read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-01-26 (Estimated); Study Completion 2024-01-26 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQOL) measured by the Severe Respiratory Insufficiency Questionnaire (SRI) | Twelve weeks
  SRI is a validated tool to assess HRQOL in patients with chronic respiratory failure receiving home mechanical ventilation, and has been shown to be applicable to different respiratory diseases. It consists of eight subscales measuring different aspects of health status with lower scores (0 to 100) indicating poorer health or higher disability.

SECONDARY OUTCOMES:
Self-reported breathlessness measured by the Modified Borg Dyspnoea Scale (MBD scale) | Twelve weeks
  The Modified Borg Dyspnoea scale measures the perceived rate of difficulty of breathing on a 0 to 10 rated numerical score, which can be used during submaximal exercise in addition. A higher score indicates higher perceived breathlessness and the aim is to compare this from baseline to the end of the study.
Excessive Daytime Sleepiness measured by the Epworth Sleepiness Score (ESS) | Twelve weeks
  The ESS is a self-administered questionnaire with 8 questions and respondents are asked to rate, on a 4 point scale (0-3), their usual chances of dosing off or falling asleep. The ESS score can range from 0 to 24 and the higher the score, the higher that person's average sleep propensity in daily life or their 'daytime sleepiness'. The aim is to compare this from baseline to the end of the study.
Mean overnight arterial oxygenation (PaO2) | Twelve weeks
  The aim to is to evaluate the efficacy of NHF regarding overnight arterial oxygenation and all participants will have overnight oximetry performed twice on nasal high flow during the study, which will be compared to their baseline off treatment.
Mean overnight transcutaneous carbon dioxide monitoring (PaCO2) | Twelve weeks
  The aim is to evaluate the efficacy of NHF regarding overnight arterial carbon dioxide monitoring and all participants will have overnight carbon dioxide monitoring performed twice on nasal high flow during the study which will be compared to their baseline off treatment.
Health Care Utilisation Questionnaire | Twelve weeks
  We will collect health resource usage by a health utilisation questionnaire based on the 10 core items of Standardised Resource Use Measure to capture core items of health resource use. from hospital admissions, to general practice and community settings, as well as home visits and medications. This will allow us to present simple cost consequence data of nasal high flow and to review how it compares from baseline to the end of the study.
Tolerability of Nasal High Flow | Twelve weeks
  Assessing tolerability of nasal high flow use.
Acceptability of Nasal High Flow | Twelve weeks
  Assessing the overall experience of using nasal high flow at home.

CONTACTS AND LOCATIONS:
Overall Officials: Swapna Mandal, MBBS,PhD, Study Chair — Chief Investigator
Locations (1):
- Royal Free Hospital, Hampstead, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All study data will be disseminated at the end of the study through appropriate publication and conference abstracts.